CLINICAL TRIAL: NCT02725294
Title: Understanding Patient Management of COPD Exacerbations
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Collaborators: VA Eastern Colorado Health Care System (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vincent S. Fan, Principal Investigator, VA Puget Sound Health Care System
Other Study IDs: 00874
Record Dates: First submitted 2016-03-28; First posted 2016-03-31 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: exacerbation; access to care; telemedicine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD patients: Veterans with COPD who are cared for at VA Puget Sound Health Care System (Seattle, WA) or VA Eastern Colorado (Denver, CO) who are at high risk for a COPD exacerbation based on an exacerbation treated with prednisone or antibiotics in the year preceding enrollment.
  Interventions: Other: This is an observational study without an intervention
- Informal Caregiver for COPD patients: Informal caregiver (ie. family member, friend, etc.) for the patient with COPD who is participating in the COPD patients cohort.
  Interventions: Other: This is an observational study without an intervention

INTERVENTIONS:
Other: This is an observational study without an intervention — Not applicable. This is an observational study without an intervention.

SUMMARY:
This observational study will examine the care-seeking behaviors of Veterans with chronic obstructive pulmonary disease (COPD) to see whether patients' perceived need for care or lack of access to care leads to delays in getting care for COPD exacerbations. Participants complete a baseline in-person visit and receive calls every two weeks for one year to monitor for COPD exacerbations. Detailed information about each exacerbation and time to care are obtained. A sample of participants and their caregivers participate in in-depth interviews. Approximately half the participants will also use a remote inhaler monitor to record their albuterol inhaler use to see if this approach can identify early exacerbations. Results from this study will be used to develop an intervention that will assist Veterans in the early identification, evaluation, and treatment of exacerbations, and will be integrated with the VA primary care team.

DETAILED DESCRIPTION:
Prompt treatment of chronic obstructive pulmonary disease (COPD) exacerbations with oral steroids and/or antibiotics, ideally within 3 days of onset of symptoms, can decrease the severity and duration of exacerbations and may reduce the risk of COPD hospitalizations. This observational study will examine Veterans' care-seeking behaviors and will focus on patients' perceived need for care and perceived access to care and whether these factors delay seeking care for COPD exacerbations, increasing the risk for hospitalizations. This study will also evaluate one approach of identifying early exacerbations through the use of a remote inhaler monitoring system.

This observational cohort study enrolled 412 Veterans with COPD at high-risk for exacerbations. As of March 2019, 246 participants have completed the 1 year follow-up; 133 are in follow-up. The Specific Aims are: 1) Examine the barriers to seeking care for COPD exacerbations or worsening breathing; 2) Test the use of a real-time remote inhaler monitor to identify early exacerbations.

All participants attended one in-person baseline visit to complete spirometry and baseline questionnaires. Participants are contacted every 2 weeks for 1 year using an interactive voice response system that screens for COPD exacerbations with 4 yes/no questions. Participants with a positive screen are called back by research staff to obtain additional detailed information on the exacerbation and how it was treated. Data analysis will examine whether access to care and baseline factors are associated with a delay in treatment.

The participants enrolled at two sites: 252 participants at VA Puget Sound in Seattle, WA and 160 participants at the VA Eastern Colorado in Denver, CO. For Aim 1, 60 participants who reported a COPD exacerbation (either hospitalized, seen in the emergency department, treated as outpatients, or did not seek treatment) participated in in-depth semi-structured interviews by a trained research staff to understand how they responded to their worsening symptoms and decided whether to seek care. 24 caregivers for these Veterans were interviewed about their perspective on the exacerbation event.

In Aim 2, 145 participants from Aim 1 used an inhaler monitor with their albuterol inhaler during the 12-month follow-up period, which transmits real-time data about their daily inhaler use. Data analysis will measure whether a change in albuterol use can predict patient reported COPD exacerbations to determine the appropriate cut-offs that can be used in a future intervention trial.

These aims will provide detailed information on how best to intervene to ensure prompt identification and treatment of COPD exacerbations. New health care delivery approaches will assist Veterans in early identification of exacerbations and provide early access to care that can be integrated into the VA primary care, emergency medicine and pulmonary specialty care settings.

ELIGIBILITY:
Veteran Cohort:

Inclusion Criteria:

1. COPD diagnosis
2. Spirometry showing FEV1/VC<0.70
3. COPD exacerbation treated with prednisone and/or antibiotics, or that resulted in a visit to the emergency department or hospitalization in the previous 12 months
4. English speaking
5. Access to telephone

Exclusion Criteria:

1. nursing home resident
2. institutionalized, imprisoned
3. life expectancy < 1 year

Informal Caregiver Cohort:

Inclusion Criteria:

1. Identified by Veteran patient as informal caregiver
2. English speaking
3. Access to telephone
4. >=18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive pulmonary disease (COPD) who receive care at the VA Puget Sound Health Care System in Seattle, WA or the VA Eastern Colorado Health Care System in Denver, CO. Informal caregivers (ie. family member or friend) to the Veteran subject will also be included
Sampling Method: Non-Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Decision to seek care | Determined for each exacerbation event during the 1-year follow-up period
  All participants with at least one exacerbation will be included in this analysis. Individuals could have both treated or untreated exacerbations and the unit of analysis will be each patient-exacerbation event. The outcome will be whether the patient sought treatment (yes/no) for their COPD exacerbation.

SECONDARY OUTCOMES:
Treatment delay | Determined for each treated exacerbation event during the 1-year follow-up period
  Only patients with ≥1 treated exacerbation during follow-up will be included in this analysis. A patient could have more than one exacerbation, and the unit of analysis will be each patient-exacerbation event

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Locke ER, Thomas RM, Simpson TL, Fortney JC, Battaglia C, Trivedi RB, Gylys-Colwell J, Swenson ER, Edelman JD, Fan VS. Cognitive and Emotional Responses to Chronic Obstructive Pulmonary Disease Exacerbations and Patterns of Care Seeking. Ann Am Thorac Soc. 2024 Apr;21(4):559-567. doi: 10.1513/AnnalsATS.202303-287OC. PMID 37966313
- [Derived] Locke ER, Young JP, Battaglia C, Simpson TL, Trivedi R, Simons C, Fortney JC, Hebert P, Swenson ER, Edelman J, Fan VS. Care-seeking and delay of care during COPD exacerbations. NPJ Prim Care Respir Med. 2022 Feb 15;32(1):7. doi: 10.1038/s41533-022-00269-9. PMID 35169140